CLINICAL TRIAL: NCT03688386
Title: Bridging Connections: A Language Intervention Study of Preterm Infants in the NICU
Brief Title: A Language Intervention Study of Preterm Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pending
Record Dates: First submitted 2018-06-18; First posted 2018-09-28 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Language Development; Language Delay; Mother-Infant Interaction; Maternal Behavior
Keywords: Language intervention; Preterm reading; Heart rate variability; Mother-infant interaction; NICU Network Neurobehavioral Scale; LENA
MeSH Terms: conditions — Language Development Disorders

STUDY DESIGN:
Intervention Model Description: Randomization of mother infant pairs to a language curriculum with reading (intervention) or an infant bonding curriculum (control)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Language Intervention (Experimental): 1. Review language and infant bonding curriculum 2. 1st LENA recording and heart rate variability of mother reading to infant 3. Provide LENA linguistic feedback and review curriculum 4. 2nd LENA recording and heart rate variability of mother reading to infant 5. Provide LENA linguistic feedback and review curriculum 6. 3rd LENA recording and heart rate variability of mother reading to infant 7. Provide LENA linguistic feedback
  Assessments: 1. NICU Network Neurobehavioral Scale (NNNS) profile at 36 weeks 2. Fragile Infant Parent Readiness Evaluation at 36 weeks 3. Parent perception survey of reading and curriculum at 36 weeks and 12 months 4. Bayley Scales of Infant and Toddler Development at 12 and 24 months 5. DNA methylation of genes pre and post intervention
  Interventions: Behavioral: Reading intervention; Behavioral: Infant bonding; Behavioral: LENA recording; Behavioral: LENA linguistic feedback
- Infant bonding (Active Comparator): 1. Review infant bonding curriculum with mother 2. 1st LENA recording and heart rate variability of mother holding infant 3. Review infant bonding curriculum 4. 2nd LENA recording and heart rate variability of mother holding infant 5. Review infant bonding curriculum 6. 3rd LENA recording and heart rate variability of mother holding infant 7. Provide linguistic feedback of all 3 LENA recordings
  Assessments: 1. NICU Network Neurobehavioral Scale (NNNS) profile at 36 weeks 2. Fragile Infant Parent Readiness Evaluation at 36 weeks 3. Parent perception survey of reading and curriculum at 36 weeks and 12 months 4. Bayley Scales of Infant and Toddler Development at 12 and 24 months 5. DNA methylation of genes pre and post intervention
  Interventions: Behavioral: Infant bonding; Behavioral: LENA recording; Behavioral: LENA summary

INTERVENTIONS:
Behavioral: Reading intervention — Written packet with 3 lessons. The first lesson includes how to begin to read and talk to their baby. The second lesson includes reading or talking about the day using parentese talk. The third lesson includes continuing to engage with the baby through interactive reading.
  Arms: Language Intervention
Behavioral: Infant bonding — Written packet with 3 lessons. The first lesson includes skin-to-skin and learning about their baby. The second lesson includes learning readiness cues and participation in feeding times. The third lesson includes developing routines and playing games.
Behavioral: LENA recording — The LENA device provide 16 hours of language recordings placed inside an infant vest. The recordings are uploaded to a computer which analyzes total adult word counts, infant vocalizations, conversational turns, background noise, and silence.
Behavioral: LENA linguistic feedback — LENA recordings of adult word counts, infant vocalizations, and conversational turns will be provided in printed form after each recording with review of each recording and progress over time.
  Arms: Language Intervention
Behavioral: LENA summary — All 3 LENA recording summaries of adult word counts, infant vocalizations, and conversational turns will be summarized in printed form and provided to mother at discharge.
  Arms: Infant bonding

SUMMARY:
This is a randomized controlled trial to study a reading intervention in the NICU among preterm infants using LENA (Language Environment Analysis) recordings, linguistic feedback, and a language curriculum to improve the neonatal inpatient language environment and language outcomes for preterm infants.

DETAILED DESCRIPTION:
This project aims to examine how an educational reading intervention in the NICU can impact preterm infant language development and examine the impact of reading on mother-infant autonomic systems. Investigators plan to determine the effects of parent reading in addition to standard caretaking and holding on preterm infants, between 23 to 31 weeks gestation hospitalized in the Women & Infants NICU, on adult word count, infant vocalizations, conversational turns through audio recording obtained over 3 separate days when the infant is corrected to 32, 34 and 36 weeks. Investigators aim to determine the effect of parent reading on maternal and infant heart rate variability before, during, and after the shared reading intervention through video and a single channel electrocardiographic recording over the same 3 separate days as the LENA recording. Additionally, investigators aim to determine the effect of parent reading on maternal stress and perceived well-being in the NICU through a validated questionnaire and to determine parent satisfaction of a NICU reading intervention through a parent questionnaire completed prior to infant discharge and at the 12 month follow up visit. Secondary outcomes include determining the effect of parent reading on infant DNA methylation of the several genes through two saliva samples collected from the infant prior to study and post study enrollment and examine its relationship with infant stress and self-regulation based on a neurobehavioral exam performed at 36 weeks corrected age. Final outcomes include examination of the long-term effect of inpatient shared reading education on infant receptive and expressive language development at 12 and 24 months. Investigators hope this research will contribute to the growing research supporting early language development in preterm infants and its impact on maternal-infant well-being.

ELIGIBILITY:
Inclusion Criteria:

* 21-31 week infants, medically stable infants, English speaking mothers over 18 years old

Exclusion Criteria:

* Intubated or medically unstable, major congenital anomalies, non English speaking

Ages: 23 Weeks to 31 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 67 (Actual)
Dates: Start 2018-12-04 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
LENA Counts | Change from 32 week language counts to 36 week language counts
  Adult word counts, conversational turns, and infant vocalizations from each recording

SECONDARY OUTCOMES:
Neonatal Intensive Care Unit Network Neurobehavioral Scale profile | 36 weeks
  A validated neurologic assessment of infant neurobehavioral, neurologic and stress responses, and regulatory capacities. The following summary scores and their minimum and maximum scores are as follows: habituation (1-9), attention (1-9), handling (0-1), quality of movement (1-3), regulation (1-9), non optimal reflexes (0-12), asymmetric reflexes (0-7), stress/abstinence (0-1), arousal (1-9), hypertonicity (0-5), hypotonicity (0-3), excitability (0-9), lethargy (0-10). Higher scores indicate the summary score, for example a higher hypertonicity score indicates increased muscle tone whereas a higher hypotonicity score indicates decreased muscle tone. Summary scores are compared to normative scores for high risk preterm infants to compare overall neurobehavior.
Bayley Scales of Infant and Toddler Development, Third Edition | 12 months and 24 months
  Individual assessment used to assess development of infants between 1 to 42 months of age. Domains and their minimum and maximum scores are as follows: adaptive behavioral (40-160), cognitive 55-145), language (47-153), motor (46-154), and social emotional (55-145). Scores can be used to assess infants progress over time.
Maternal Well-Being | 36 weeks
  Using the Fragile Infant Parent Readiness Evaluation survey to evaluate maternal well-being
Perception of reading and infant bonding | 36 weeks and 12 months
  Parent survey regarding her experience in the NICU with reading, curriculum, and future plans to read to her infant

OTHER OUTCOMES:
DNA methylation | Enrollment and 36 weeks
  Understand DNA methylation pattern differences of genes of before and after study participation.

CONTACTS AND LOCATIONS:
Overall Officials: Betty Vohr, MD, Principal Investigator — Women and Infants Hospital of Rhode Island
Locations (1):
- Women and Infants Hospital of Rhode Island, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Feldman R, Magori-Cohen R, Galili G, Singer M, Louzoun Y. Mother and infant coordinate heart rhythms through episodes of interaction synchrony. Infant Behav Dev. 2011 Dec;34(4):569-77. doi: 10.1016/j.infbeh.2011.06.008. Epub 2011 Jul 20. PMID 21767879
- [Background] Lester BM, Marsit CJ, Giarraputo J, Hawes K, LaGasse LL, Padbury JF. Neurobehavior related to epigenetic differences in preterm infants. Epigenomics. 2015 Oct;7(7):1123-36. doi: 10.2217/epi.15.63. Epub 2015 Nov 20. PMID 26585459
- [Background] Lariviere J, Rennick JE. Parent picture-book reading to infants in the neonatal intensive care unit as an intervention supporting parent-infant interaction and later book reading. J Dev Behav Pediatr. 2011 Feb-Mar;32(2):146-52. doi: 10.1097/DBP.0b013e318203e3a1. PMID 21289497
- [Result] Caskey M, Stephens B, Tucker R, Vohr B. Adult talk in the NICU with preterm infants and developmental outcomes. Pediatrics. 2014 Mar;133(3):e578-84. doi: 10.1542/peds.2013-0104. Epub 2014 Feb 10. PMID 24515512